CLINICAL TRIAL: NCT03504878
Title: Cost-effectiveness Analysis and Case-based Payment Norm Modeling on Appendicitis Patients at Hanoi Medical University Hospital
Status: Completed | Type: Observational
Sponsor: Hanoi Medical University (Other)
Responsible Party: Principal Investigator, Bui My Hanh, Director, Science Research and International Cooperation Unit, Hanoi Medical University
Other Study IDs: HMU16224
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2018-04-20 (Actual); Status verified 2018-04

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients undergoing laparoscopic appendectomy: Appendix removal via scope.
  Interventions: Procedure: Laparoscopic appendectomy
- Patients undergoing open appendectomy: Open operation for removal of appendix
  Interventions: Procedure: Open appendectomy

INTERVENTIONS:
Procedure: Laparoscopic appendectomy — The laparoscopic appendectomy was performed with three trocars. Pneumoperitoneum was created using an open Hasson technique. The mesoappendix was divided using a harmonic scalpel or endoscopic tissue fusion device. The appendix was divided by placing one endoscopic loop and cut with harmonic scalpel. The specimen was removed through the umbilical port.
  Groups: Patients undergoing laparoscopic appendectomy
Procedure: Open appendectomy — The open appendectomy was carried out in the standard way with McBurney muscle splitting incision.
  Groups: Patients undergoing open appendectomy

SUMMARY:
In the world, there are several studies comparing the cost-effectiveness between laparoscopic appendectomy and open appendectomy. But in Vietnam, health economics studies for acute appendicitis surgery in general and laparoscopic appendectomy in particular has hardly been available, and in the context of reform of the financial mechanism for payment, questions about the cost-effectiveness between the two surgical methods are particularly concerned. Therefore, we conducted a study "Cost-effectiveness analysis and case-based payment norm modeling in patients with appendectomy at Hanoi Medical University Hospital"

DETAILED DESCRIPTION:
Acute Appendicitis (AA) is a surgical emergency most common stomach. Appendicitis occurs at all ages. Recently, the rate tends to increase VRTC with age. In the United States, there are about 300,000 cases of appendectomy surgery per year. In Vietnam, according to statistics from a number of other authors showed that the rate of appendectomy surgery accounted for 40.5% - 49.8% of total number of cases of abdominal emergency. Open appendectomy (OA) has long been applied as the gold standard surgical procedure for the treatment of AA for over a century, since it was introduce by McBurrney in 1894 and still be common choice for procedure in many center. In 1981, due to the growth of endoscopic surgery, Semm first introduced the laparoscopic appendectomy, which render a minimal invasive procedure for abdomen and skin, nevertheless, its superiority over open appendectomy (OA) is still being debated. Some more recent paper demonstrate that Laparoscopic Appendectomy is the technique of choice in treatment of AA because of its clinical advantage and cost-effectiveness, however, more than 20 years later, the benefits of LA still remain a controversy for many researchers.

There are several studies comparing the cost-effectiveness between laparoscopic appendectomy and open appendectomy in the world. But in Vietnam, health economics studies for appendix removal surgery in general and laparoscopic appendectomy in particular has hardly been available, and in the context of reform of the financial mechanism for payment, questions about the cost-effectiveness between the two surgical methods are particularly concerned. Therefore, we conducted a study "Cost-effectiveness analysis and case-based payment norm modeling in patients with appendectomy at Hanoi Medical University Hospital" with two main purposes

1. Analyze cost-effectiveness between laparoscopic and open surgery in patients undergoing appendectomy at Hanoi Medical University Hospital in 2011 - 2013
2. Model case-based payment norm of appendectomy patients at Hanoi Medical University Hospital

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic Appendectomy patients agree to participate in research and are paid by the mode of service charge
* Laparoscopic Appendectomy patients agree to participate in research and are paid according to package medical cases

Exclusion Criteria:

* Patients with combined pathology affecting surgical outcomes
* The patient did not agree to participate in research
* Patients do not comply with treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with clinical, laboratory, and radiological signs of acute appendicitis
Sampling Method: Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Average cost of hospitalization based on the final hospital bills | 2 years
  Total mean expense that patient pay for hospital after completing acute appendicitis treatment
Average Cost of medication | 2 years
  Total mean cost of drugs used during operation for removal of appendix
Overall treatment cost of acute appendicitis patient | From the beginning of hospital admission till discharge from hospital ((an expected average of 10 days, maximum 20 days)
  Total amount of money that acute appendicitis patient have to spend during the time of hospitalization
Case-based cost of appendectomy | 2 years
  The expenses that patient pay for surgical removal of appendix accounted by case-based standardisation
Cost of appendectomy based on health care services fee | 2 years
  The expenses that patient pay for acute appendicitis treatment accounted in accordance with services fee of hospital

SECONDARY OUTCOMES:
Length of hospital stay | from the beginning of the surgery till discharge from hospital (an expected average of 8 days, maximum 20 days)
  No. of days from surgery to discharge of hospital
Duration of post-operative pain | from the beginning of the surgery till discharge from hospital (an expected average of 8 days, maximum 20 days)
  No. of days that patient experience pain after surgery
Degree of post-operative pain | from the beginning of the surgery till discharge from hospital (an expected average of 8 days, maximum 20 days)
  Percentage of patients according to stratification of post-operative pain
Time until resumption of clear liquid and regular diet | from the beginning of the surgery to the resumption (an expected average 2 days after the surgery
  No. of days from surgery to the resumption of clear liquid and regular diet
Surgical outcome at hospital discharge | 2 years
  Percentage of patients with good outcome at hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code